CLINICAL TRIAL: NCT01078207
Title: A Prospective Non-Randomized Study of Pulse Oximetry Saturation Patterns in Postoperative Patients at High Risk of Obstructive Sleep Apnea
Brief Title: Oxygen Saturation Patterns in Post-Op Patients at Risk for Obstructive Sleep Apnea
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: COV-MO-PO-A105
Record Dates: First submitted 2010-02-26; First posted 2010-03-02 (Estimated); Results first posted 2012-08-01 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study will include patients who have major surgery and are at risk for or have been diagnosed with sleep apnea. The patients will be monitored the night after surgery for repeating episodes of reduced breathing and oxygen levels. The study will determine if episodes of decreased breathing are reflected in the oxygen monitor.

DETAILED DESCRIPTION:
There is no further detailed description available.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years undergoing thoracic, vascular, head and neck, gynecological, urological, general, orthopedic, and plastic surgery.
* Patient must require analgesia and/or sedation postoperatively by any route (intravenous, intramuscular, oral, epidural or intrathecal) for the duration of the study
* Postoperative patients with at least one anticipated over night stay on the general ward with a minimum length of 14 hrs.
* Patients in the ASA category 1-4
* Patients at high risk for obstructive sleep apnea (OSA) as identified by the STOP-Bang Questionnaire or patients previously diagnosed with OSA and not using a CPAP device. (No screening with STOP needed for these patients.)
* Spontaneous breathing

Exclusion Criteria:

* Age less than 18 years
* Patients receiving or anticipated to receive postoperative positive airway pressure support
* Previous allergic/contact reactions to adhesives
* Patients unable to give informed consent
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years undergoing thoracic, vascular, head and neck, gynecological, urological, general, orthopedic, and plastic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Mecca, MD, Study Chair — Medtronic - MITG
Locations (2):
- Canada (2):
  - Toronto General Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From Feb 2010 to Oct 2010 adults at high risk for obstructive sleep apnea scheduled for general surgery requiring analgesia with an expected over night hospital stay were recruited from the hospital clinic.
Groups:
- Adult Surgical Patients At Risk for Obstructive Sleep Apnea: Observational study of adult patients at high risk for obstructive sleep apnea undergoing general surgery requiring analgesia with an expected over night stay. All patients were in this group.
Period: Overall Study
Arm/Group | Adult Surgical Patients At Risk for Obstructive Sleep Apnea
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Adult Surgical Patients At Risk for Obstructive Sleep Apnea
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 51
  >=65 years | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 78
Region of Enrollment [Number; unit: participants]
  Canada | 100

OUTCOME MEASURES:

1. Primary Outcome: Presence of Repetitive Reductions in Nasal Airflow Patterns in the Pulse Oximetry Saturation Trend Data.
Description: Number of patients exhibiting the presence of repetitive reductions in airflow patterns in the pulse oximetry trend data collected on subjects
Time Frame: 12 hour after released from the recovery room
Population: All patients with complete data were analyzed.
Measure: Number; unit: participants
Arm/Group | Adult Surgical Patients At Risk for Obstructive Sleep Apnea
Number analyzed (Participants) | 83
participants | 30

2. Secondary Outcome: Relationship Between the Oxygen Desaturation Patterns and Repetitive Reductions in Nasal Airflow as Measured by Inductance Plethysmography and Nasal Pressure.
Description: The number of patients with a positive repetitive reduction in nasal airflow which correlates with positive oxygen desaturation pattern as measured by photoplethysmography sensors.
Time Frame: 12 hours after discharge form the recovery room
Population: All patients with a positive repetitive reduction in nasal airflow.
Measure: Number; unit: participants
Arm/Group | Adult Surgical Patients At Risk for Obstructive Sleep Apnea
Number analyzed (Participants) | 30
participants | 20

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Adult Surgical Patients At Risk for Obstructive Sleep Apnea
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less